CLINICAL TRIAL: NCT05182580
Title: Assessing the Impact of Using Autonomous Artificial Intelligence (AI) for Pre-screening of Diabetic Retinopathy (DR) and Diabetic Macular Edema on Physician Productivity in Bangladesh
Brief Title: Bangladesh PRODUCTIVity in Eyecare Trial
Acronym: B-PRODUCTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orbis (Other)
Collaborators: Digital Diagnostics, Inc. (Industry); Deep Eye Care Foundation (DECF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: ORBIS-DXS-DECF-2021
Record Dates: First submitted 2021-11-16; First posted 2022-01-10 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Intervention Model Description: Cluster-randomized (by clinic day) controlled trial.
Who Masked: Participant, Care Provider
Masking Description: The retina specialists are masked both to patient group assignment (that is, whether autonomous AI results were used or not on the particular clinic day) and also masked to the results of the autonomous AI on Intervention days. Patients are also masked to group assignment and autonomous AI screening results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Group (Experimental): Autonomous AI results are used to evaluate if the participant needs to see the retina specialist (positive result) or not (negative result).
  Interventions: Diagnostic Test: Results utilized from autonomous AI diagnostic system for diabetic retinopathy and/or diabetic macular edema
- Control Group (No Intervention): All participants see the retina specialist irrespective of the results of their autonomous AI evaluation.

INTERVENTIONS:
Diagnostic Test: Results utilized from autonomous AI diagnostic system for diabetic retinopathy and/or diabetic macular edema — If patients receive a negative result they do not see the retina specialist
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to assess the impact of using autonomous artificial intelligence (AI) system for identification of diabetic retinopathy (DR) and diabetic macular edema on productivity of retina specialists in Bangladesh.

Globally, the number of people with diabetes mellitus is increasing. Diabetic retinopathy is a chronic, progressive complication of diabetes mellitus that affects the microvasculature of the retina, which if left untreated can potentially result in vision loss. Early detection and treatment of diabetic retinopathy can prevent potential blindness.

Study Aim: To assess the impact of using autonomous artificial intelligence (AI) system for detection of diabetic retinopathy (DR) and diabetic macular edema on physician productivity in Bangladesh.

Main study question: Will ophthalmologists with clinic days randomized to use autonomous AI DR detection for all persons with diabetes (diagnosed or un-diagnosed) visiting their clinic system have a greater number of examined patients with diabetes (by either AI or clinical exam), and a greater complexity of examined patients on a recognized grading scale, per physician working hour than those randomized not to have autonomous AI screening for their diabetes population?

The investigators anticipate that this study will demonstrate an increase in physician productivity, supporting efficiency for both physicians and patients, while also addressing increased access for DR screening; ultimately, preventing vision loss amongst diabetic patients. The study has the potential to contribute to the evidence base on the benefits of AI for physicians and patients. Additionally, the study has the potential to demonstrate the benefits (and/or challenges) of implementing AI in resource-constrained settings, such as Bangladesh.

DETAILED DESCRIPTION:
Bangladesh PRODUCTIVity in Eyecare (B-PRODUCTIVE) Trial

Study Aim: To assess the impact of using autonomous artificial intelligence (AI) for identification of diabetic retinopathy (DR) and diabetic macular edema on productivity of retina specialists in Bangladesh.

Hypothesis: Autonomous AI increases retina specialist productivity

Main Study Question: Will retina specialists complete a greater number of diabetic eye exams per working hour (including persons reviewed by AI whom the retina specialist does not need to see personally) when they use autonomous AI in a randomized clinical trial?

Design: Cluster-randomized (by clinic day) controlled trial.

Randomization: By clinic day. Each morning the clinic manager will open an opaque envelope, which informs the manager if it is an Intervention (AI) or Control (non-AI) day.

Interventions: All patients in both groups go through the eligibility checklist. If approved, they will be evaluated by autonomous AI. This is done to decrease potential bias (neither patients nor physicians know the group assignment of participants) and concealment (so that neither patients nor doctors can arrange visits on a known "Intervention Day").

Intervention Group: On randomly selected "Intervention" clinic days, if patients screen positive or have insufficient image quality, they continue to the ophthalmologist. If not eligible for autonomous AI, they proceed straight to the ophthalmologist without autonomous AI evaluation. If patients receive a negative result, they do not see the retina specialist, and are referred for a visit at the regular eye clinic (not the retina clinic) in 3 months.

Control Group: On randomly-selected "Control Days," all patients see the ophthalmologist, irrespective of the results of autonomous AI evaluation.

Masking: The retina doctors are masked both patient group assignment (that is, whether autonomous AI was used for pre-screening or not on the particular clinic day) and also masked to the results of the AI on Intervention days. Patients are also masked to group assignment and autonomous AI results.

ELIGIBILITY:
Inclusion Criteria:

Retina specialists regularly seeing patients with DR

* Routinely examines >= 20 patients with diabetes without known diabetic retinopathy or diabetic macular edema per week
* Routinely provides laser treatment or intravitreal injections to >= 3 DR patients/month

Patients

* Diagnosed with type 1 or 2 diabetes
* Presenting visual acuity >= 6/18 best corrected visual acuity in the better-seeing eye

Exclusion Criteria:

Retina specialists

* Currently using an AI system integrated into their clinical care and/or inability to provide informed consent.

Patients

* Inability to provide informed consent or understand the study; persistent vision loss, blurred vision or floaters; previously diagnosed with diabetic retinopathy or diabetic macular edema; history of laser treatment of the retina or injections into either eye, or any history of retinal surgery; contraindicated for imaging by fundus imaging systems

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 993 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, MD, MPH, Study Chair — Orbis
Locations (1):
- Deep Eye Care Foundation, Rangpur City, Bangladesh

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD

REFERENCES:
- [Derived] Abramoff MD, Whitestone N, Patnaik JL, Rich E, Ahmed M, Husain L, Hassan MY, Tanjil MSH, Weitzman D, Dai T, Wagner BD, Cherwek DH, Congdon N, Islam K. Autonomous artificial intelligence increases real-world specialist clinic productivity in a cluster-randomized trial. NPJ Digit Med. 2023 Oct 4;6(1):184. doi: 10.1038/s41746-023-00931-7. PMID 37794054

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The random allocation of each cluster (clinic day) was concealed until clinic staff received an email with this information just before the start of that day's clinic. Medical staff who determined access, specialists and patient participants remained masked to the random assignment of clinic days as control or intervention. Technicians and/or specialists are not considered enrolled. The participant flow details patient participants randomized by clinic day.
Units Other Than Participants: clinic days
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 494; 51 clinic days (Patient participants randomized by clinic day) | 499; 54 clinic days (Patient participants randomized by clinic day)
Completed | 494; 51 clinic days | 499; 54 clinic days
Not Completed | 0; 0 clinic days | 0; 0 clinic days

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 494 | 499 | 993
Age, Customized [Mean (Standard Deviation); unit: years]
  Age, years | 50.8 (9.70) | 51.0 (10.0) | 50.9 (9.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 265 | 524
  Male | 235 | 234 | 469
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Bangladesh | 494 | 499 | 993

OUTCOME MEASURES:

1. Primary Outcome: Number of Completed Care Encounters Among Clinic Patients With Diabetes Per Retina Specialist Clinic Hour
Description: Number of completed care encounters among clinic patients with diabetes per retina specialist clinic hour. Numerator is the number of care encounters among patients with diabetes (including persons evaluated by autonomous AI on Intervention Days who are determined not to need to see the retina specialist). The denominator is retina specialist clinic time in hours.
Time Frame: 105 randomized clinic days
Population: Completed care encounters among clinic patients with diabetes
Measure: Mean (95% Confidence Interval); unit: care encounters/specialist clinic hour
Units Other Than Participants: care encounters pts with diabetes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 494 | 499
Number analyzed (care encounters pts with diabetes) | 1189 | 920
care encounters/specialist clinic hour | 1.59 [1.3 to 1.8] | 1.14 [1.02 to 1.25]

2. Primary Outcome: Number of Completed Care Encounters Among All Clinic Patients (With and Without Diabetes) Per Retina Specialist Clinic Hour
Description: Number of completed care encounters among all clinic patients (with and without diabetes) per retina specialist clinic hour. Numerator is the number of completed care encounters (including persons evaluated by autonomous AI on Intervention Days who are determined not to need to see the retina specialist). The denominator is retina specialist clinic working time in hours.
Time Frame: 105 randomized clinic days
Population: All retina clinic care encounters
Measure: Mean (95% Confidence Interval); unit: care encounters/specialist clinic hour
Units Other Than Participants: all retina clinic care encounters
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 494 | 499
Number analyzed (all retina clinic care encounters) | 3014 | 2708
care encounters/specialist clinic hour | 4.05 [3.66 to 4.43] | 3.36 [3.08 to 3.63]

3. Secondary Outcome: Specialist Productivity Adjusted for Patient Complexity for Patients With Diabetes
Description: Specialist productivity (care encounters / specialist clinic hour) adjusted for patient complexity for patients with diabetes.
  The complexity score for each patient participant was calculated by a masked United Kingdom National Health Service grader using the International Grading system, adapted from Wilkinson et al. International Clinical Diabetic Retinopathy and Diabetic Macular Edema Severity Scales (no DED = 0 points, mild non-proliferative DED = 0 points, moderate or severe non-proliferative DED = 1 point, proliferative DED = 3 points and diabetic macular edema = 2 points.) The patient participant complexity score was summed across both eyes. The average complexity score for each arm was calculated.
  Complexity adjusted specialist productivity was calculated for intervention and control arms by multiplying the respective overall productivity (care encounters per specialist clinic hour) calculation by the respective average complexity score.
Time Frame: 105 randomized clinic days
Population: This is the same calculation as Outcome 1 but with the addition of adjustment for complexity.
  (# retina care encounters*complexity score) / specialist clinic hours
Measure: Number; unit: (exams/clinic hour)*(score on a scale)
Units Other Than Participants: care encounters pts with diabetes
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 494 | 499
Number analyzed (care encounters pts with diabetes) | 1189 | 920
(exams/clinic hour)*(score on a scale) | 3.15 | 1.19

4. Secondary Outcome: Number of Participants Who Were Very Satisfied or Satisfied With Autonomous AI
Description: After the patient participant completed the autonomous AI process, a survey with a 4-point Likert scale ("very satisfied," "satisfied," "dissatisfied," "very dissatisfied") was administered, concerning the participant's satisfaction with interactions with the healthcare team, time to receive examination results, and receiving their diagnosis from the autonomous AI system.
Time Frame: 105 randomized clinic days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 494 | 499
Participants | 493 | 499

ADVERSE EVENTS:
Time Frame: Through study completion, up to 5 months
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/494 | 0/499
Serious Adverse Events (participants affected / at risk) | 0/494 | 0/499
Other Adverse Events (participants affected / at risk) | 0/494 | 0/499

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT05182580/Prot_SAP_000.pdf